CLINICAL TRIAL: NCT04356183
Title: Weight Loss and Exercise To Improve Rheumatoid Arthritis Cardiovascular Risk
Acronym: SWET/CHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00104843; R21AR076663 (NIH)
Record Dates: First submitted 2020-04-13; First posted 2020-04-22 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: RA Seropositive; RA Erosive; Exercise; Diet; Nutrition; Cardiovascular Risk
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling Health As Treatment (CHAT) (Other): CHAT is a control arm designed to reflect traditional clinical counselling.
  Interventions: Other: CHAT: Counseling Health As Treatment
- Supervised Weight loss and Exercise Training (SWET) (Experimental): SWET includes supervised aerobic (3x/w) and resistance (2x/w) training plus a weekly weight loss session.
  Interventions: Other: SWET: Supervised Weight loss and Exercise Training

INTERVENTIONS:
Other: SWET: Supervised Weight loss and Exercise Training — Weight loss will occur via a dietitian-led intervention targeting weight loss over 16 weeks, with weekly weigh-ins and group support sessions. Exercise training will consist of three times per week of an interval-based aerobic program plus twice-weekly resistance training. Both weight loss and exercise training will be supervised to maximize safety and adherence.
  Arms: Supervised Weight loss and Exercise Training (SWET)
Other: CHAT: Counseling Health As Treatment — Control Arm over 16 weeks.
  Arms: Counseling Health As Treatment (CHAT)

SUMMARY:
This is a small exploratory, randomized, controlled trial. Twenty-six older (ages 60-80 yr.), obese (BMI 28-40 kg/m2) persons with rheumatoid arthritis (RA) (seropositive or erosive) will be randomized to 16 weeks of a counseling health as treatment (CHAT) program or a supervised weight loss and exercise training (SWET) program.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 28-40 kg/m2.
* Must have internet access.
* Seropositive (positive rheumatoid factor or anti-citrullinated protein antibody) or erosions typical of RA on radiographs.

Exclusion Criteria:

* Subject unwilling/unable to utilize online platforms (e.g. ZOOM, REDCap, Pattern Health) for study activities.
* Current use of biologic agents other than those targeting tumor necrosis factor alpha.
* Current (within the last month) pharmacologic therapy with corticosteroids at doses greater than prednisone 5mg per day (or equivalent glucocorticoid doses).
* Participating in regular exercise within the past 3 months (According to 2018 US guidelines: Not more than 150 minutes per week of moderate intensity exercise or 75 minutes per week of vigorous intensity exercise).
* New medications within the last three months and stable doses for ≥ 1 month.
* Diagnosis of coronary artery disease.
* Diagnosis of type 2 diabetes mellitus.
* Other inflammatory arthropathy or myopathy, Paget's disease, pigmented villonodular synovitis, joint infection, ochronosis, neuropathic arthropathy, osteochondromatosis, acromegaly, hemochromatosis, or Wilson's disease.
* Absolute contra-indications to exercise: Recent (<6 months) acute cardiac event, unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurism or acute systemic infection.
* Relative contra-indications to exercise: Left main coronary stenosis, moderate stenotic valvular heart disease, outflow tract obstruction, high degree AV block, ventricular aneurysm, uncontrolled metabolic disease (e.g. diabetes, thyrotoxicosis, myxedema), uncontrolled pulmonary disease (e.g. severe COPD or pulmonary fibrosis), mental or physical impairment leading to inability to exercise adequately.
* Significant weight change (gain or loss of > 10 pounds in 1 month) within the past 6 months.
* Unwillingness or inability to adhere to the diet structure of the study.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim G, Ross LM, Sudnick AM, Johnson JL, Pieper CF, Connelly MA, Ilkayeva O, Muehlbauer MJ, Bales CW, Porter Starr KN, Kraus WE, Andonian BJ, Huffman KM. The impact of lifestyle modification on metabolic pathways in older adults with overweight/obesity and rheumatoid arthritis: a secondary exploratory analysis of the SWET-RA study. BMC Rheumatol. 2025 Jun 9;9(1):68. doi: 10.1186/s41927-025-00525-8. PMID 40490834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were primarily recruited from outpatient rheumatology clinics serving Duke Health in North Carolina, USA. Additional recruitment strategies included: paper and electronic advertisements, physician referrals, and the Duke Health and Exercise Research registry.
Pre-assignment Details: Of the 26 consented participants, 24 participants met inclusion criteria and were randomized.
Period: Overall Study
Arm/Group | Counseling Health As Treatment (CHAT) | Supervised Weight Loss and Exercise Training (SWET)
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counseling Health As Treatment (CHAT) | Supervised Weight Loss and Exercise Training (SWET) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (6.2) | 68.1 (5.8) | 67.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Syndrome Severity Z-score (MSSc)
Description: The primary objective is to compare change in metabolic syndrome z-score (MSSc) between groups. The MSSc is a continuous weighted score of the five metabolic syndrome variables-fasting high-density lipoprotein cholesterol, triglycerides, glucose, waist circumference, and mean arterial blood pressure. A modified z-score was calculated for each participant using continuous differences between the Adult Treatment Panel (ATP) III guideline values and participant values with normalization to the cohort's standard deviations. To account for variations in ATP III criteria between men and women, the investigators used sex-specific MSSc equations. A lower MSSc indicates a better outcome.
Time Frame: Baseline and 16 weeks
Population: One SWET participant was excluded from analysis due to prior chronic lymphocytic leukemia diagnosis.
Measure: Mean (Standard Deviation); unit: Z-score (unitless)
Arm/Group | Counseling Health As Treatment (CHAT) | Supervised Weight Loss and Exercise Training (SWET)
Number analyzed (Participants) | 10 | 10
Z-score (unitless)
  Baseline | -1.89 (2.39) | -1.82 (2.01)
  Week 16 | -3.23 (2.80) | -3.49 (2.28)
Statistical Analysis 1: Comparison: Counseling Health As Treatment (CHAT) vs Supervised Weight Loss and Exercise Training (SWET); Test type: Superiority; p < 0.05, Regression, Linear

2. Secondary Outcome: Physical Function as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System) Questionnaire
Description: Change in patient-reported outcomes using PROMIS Physical Function Questionnaire. The questionnaire was scored using "response pattern scoring" according to the PROMIS scoring manual in order to calculate the T-score for this outcome measure. The population mean T-score for Physical Function is 50, with a score of 40 considered below average and a score of 60 considered above average.
Time Frame: Baseline and 16 weeks
Population: One SWET participant was excluded from analysis due to prior chronic lymphocytic leukemia diagnosis.
Measure: Mean (Standard Deviation); unit: T-score (unitless)
Arm/Group | Counseling Health As Treatment (CHAT) | Supervised Weight Loss and Exercise Training (SWET)
Number analyzed (Participants) | 10 | 10
T-score (unitless)
  Baseline | 41.7 (5.0) | 42.3 (6.3)
  16 weeks | 41.7 (6.4) | 48.1 (6.5)
Statistical Analysis 1: Comparison: Counseling Health As Treatment (CHAT) vs Supervised Weight Loss and Exercise Training (SWET); Test type: Superiority; p < 0.05, Regression, Linear

3. Secondary Outcome: Disease Activity Score (DAS-28)
Description: Change in disease activity measured using the DAS-28. DAS-28 is a composite measure including a self-reported overall health assessment on a 100 mm visual analog scale, the number of tender and swollen joints determined from a 28-joint examination, and C-reactive protein. Scores range from 0 [very well] to 10 [very poor].
Time Frame: Baseline and 16 weeks
Population: One SWET participant was excluded from analysis due to prior chronic lymphocytic leukemia diagnosis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Counseling Health As Treatment (CHAT) | Supervised Weight Loss and Exercise Training (SWET)
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 3.1 (1.0) | 2.9 (1.2)
  Week 16 | 2.9 (0.8) | 2.1 (0.9)
Statistical Analysis 1: Comparison: Counseling Health As Treatment (CHAT) vs Supervised Weight Loss and Exercise Training (SWET); Test type: Superiority; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Counseling Health As Treatment (CHAT) | Supervised Weight Loss and Exercise Training (SWET)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Counseling Health As Treatment (CHAT) (N=12) | Supervised Weight Loss and Exercise Training (SWET) (N=12)
Joint and/or muscle pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Infection (Infections and infestations) | 1 | 5
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT04356183/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT04356183/ICF_000.pdf